CLINICAL TRIAL: NCT06477692
Title: INVERT - Prospective Phase II Randomized Trial of Involved Nodal Versus Elective Neck RadioTherapy
Brief Title: Invert-Prospective Phase II Randomized Trial of Involved Nodal Versus Elective Neck RadioTherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Sher, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2024-0603; 1R01CA251792-01A1 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Drug Therapy; Cisplatin; Cetuximab

STUDY DESIGN:
Intervention Model Description: radiation ENI versus INRT
Who Masked: Participant
Masking Description: Patients are blinded to their treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard radiotherapy with elective neck irradiation (ENI) (Active Comparator): The elective neck dose is 56 Gy in 35 fractions Lymph nodes measuring 17 mm or greater in any dimension, or showing FDG above adjacent blood pool, may receive 63 Gy in 35 fractions per physician discretion.The elective neck field is determined by the primary site.
  The Oropharynx:
  Node-positive side: Levels IB-V and RP nodes Node-negative side: Levels II-IV, RP at discretion of physician For ipsilateral tonsil decision-making, see 4.1.1.6.3
  The Larynx:
  Node-positive side: Levels IB-V Node-negative side: Levels II-IV Subglottic extension: Level VI
  Hypopharynx:
  Node-positive side: Levels IB-V and RP nodes Node-negative side: Levels II-V and RP nodes Pyriform sinus involvement: Level VI
  Interventions: Drug: ENI using IMRT with or without chemotherapy; Radiation: ENI
- Involved and suspicious lymph node delineation and targeting (Experimental): After the involved and suspicious nodes are contoured, the physician will contour remaining nodes that are present on more than one CT slice and submit them to the AI-Radiomics module for assessment.The nodal gross tumor volume (GTVn, GTVns and GTVnps for involved, suspicious nodes or potentially suspicious) will be contoured on the planning CT, using radiographic and clinical information to define its extent. The total dose for GTVns is 63 Gy in 35 fractions, and the total dose for GTVnps is 56 Gy in 35 fractions. For lymph nodes identified as potentially suspicious by the AI- Radiomics module that are outside of the expected primary draining zone, physicians may not treat the lymph node if the module assesses its estimation uncertainty as greater than 50%.
  Interventions: Drug: ENI using IMRT with or without chemotherapy; Radiation: INRT

INTERVENTIONS:
Drug: ENI using IMRT with or without chemotherapy — This study is a phase II single-blinded randomized trial comparing standard ENI with involved nodal radiotherapy. INRT using intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin- paclitaxel)
  Other Names: cisplatin, cetuximab, or carboplatin- paclitaxel)
Radiation: INRT — INRT using intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin- paclitaxel)
  Arms: Involved and suspicious lymph node delineation and targeting
Radiation: ENI — ENI using IMRT with or without chemotherapy
  Arms: Standard radiotherapy with elective neck irradiation (ENI)

SUMMARY:
To determine the risk of solitary elective volume recurrence following involved nodal radiotherapy (INRT) versus elective nodal irradiation (ENI)

DETAILED DESCRIPTION:
Patients are assigned to either elective nodal irradiation (ENI), the current treatment paradigm, or involved nodal radiotherapy (INRT), the experimental treatment. INRT is more specifically targeting potentially cancerous nodes, identified using an AI program developed in-house. The hope is that this more specific targeting will decrease healthy tissue being irradiated, therefore decreasing potential side effects of the radiation treatment.

Patients are blinded during study participation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-proven diagnosis of squamous cell carcinoma of the oropharynx, larynx, or hypopharynx. Squamous cell carcinoma of unknown primary is not allowed.
* Patients must have clinically or radiographically evident measureable disease at the primary site and/or nodal stations. Diagnostic lymph node excision (≤ 2 nodes) is also allowable.
* Patients may undergo a diagnostic or therapeutic transoral resection for a T1-2 tonsil or base of tongue cancer.
* Clinical stage I-IVB (AJCC, 7th edition); stages I-II glottic cancer are excluded
* Age ≥ 18 years.
* ECOG Performance Status 0-2
* All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Neck CT and/or neck MRI, and PET-CT
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Distant metastasis.
* Inability to undergo either a diagnostic CT with contrast or simulation CT with contrast.
* Inability to undergo PET-CT.
* Stage I and II glottic carcinoma.
* Gross total excision of both the primary and nodal disease.
* Synchronous non-skin cancer primaries outside of the oropharynx, larynx, and hypopharynx except for low- and intermediate-risk prostate cancer and synchronous well-differentiated thyroid cancer; in the latter case, surgery may occur before or after treatment, provided all other eligibility criteria are met.
* Prior invasive malignancy with an expected disease-free interval of less than 3 years.
* Prior systemic chemotherapy for the study cancer; prior chemotherapy for a remote cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields.
* Subjects may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy agents in this study (if necessary).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* History of severe immunosuppression, including HIV, and organ or autologous or allogeneic stem cell transplant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
The probability at two years: SEVR in INRT versus ENI patients | 2 years
  The probability at two years will be compared between the arms using a one- sided Fisher's exact test (probability of SEVR between the arms).

SECONDARY OUTCOMES:
Incidence of Acute Grade 2+ Dermatitis between ENI vs INRT arms | Start of RT through 90 days post RT
  Comparison of instances of grade 2+ acute dermatitis between patients treated with INRT (involved nodal radiotherapy, study treatment) vs ENI (elective nodal irradiation, standard of care). This will be compared between the arms using a Fisher exact test (2-sided).
Incidence of Grade 3+ Dysphagia between ENI vs INRT arms | 2 years post RT
  Comparison of instances of grade 3+ dysphagia between patients treated with INRT (involved nodal radiotherapy, study treatment) vs ENI (elective nodal irradiation, standard of care). This will be compared between the arms using a Fisher exact test (2-sided).
MDADI Quality of Life composite score | 2 years post RT
  Comparison of MDADI composite scores at 2 years post RT between patients treated with INRT (involved nodal radiotherapy, study treatment) vs ENI (elective nodal irradiation, standard of care). Patients with disease recurrence will be excluded from analysis. At two years, both scores will be compared between the arms using a two-sided T test.

CONTACTS AND LOCATIONS:
Overall Officials: David Sher, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No